CLINICAL TRIAL: NCT01997528
Title: Efficiency of Gas Exchange Using a Miniaturized Pump Driven Veno-venous Extracorporeal Gas Exchange Device (ILA-Activve)
Brief Title: Gas Transfer on ILA-Activve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Staudinger, Ao. Univ.-Prof. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK Nr. 1191/2013
Record Dates: First submitted 2013-11-07; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Hypercapnia
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Extracorporeal CO2 elimination by ILA Activve(R) (Experimental)
  Interventions: Device: Change of blood flow or sweep gas flow ( ILA Activve)

INTERVENTIONS:
Device: Change of blood flow or sweep gas flow ( ILA Activve)

SUMMARY:
Oxygenatuion and decarboxylation during different settings (steps of blood flow and sweep gas flow) of extracorporeal gas exchange by ILA Activve using a jugular 22French double lumen cannula are measured.

ELIGIBILITY:
Inclusion Criteria:

* Patient on ILA Activve
* Controlled mechanical ventilation
* No spontaneous breathing

Exclusion Criteria:

- Pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Blood gas analysis | Changes after every 15 min. of each setting (13 settings leading to 195 min. altogether)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Staudinger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Dept. of Medicine I, ICU, General Hospital of Vienna, Vienna, Vienna, Austria